CLINICAL TRIAL: NCT01163227
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over, Single-dose Study to Evaluate the Effects of AQW051 on Cognitive Function in Patients With Chronic Stable Schizophrenia Including a One Week Multiple-dose Extension to Assess the Persistence of Observed Effects and a Multiple-dose Cross Over Study in Non Smokers Only.
Brief Title: Effect of AQW051 on Cognitive Function in Patients With Chronic Stable Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A2205
Record Dates: First submitted 2010-07-12; First posted 2010-07-15 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2013-03

CONDITIONS: Schizophrenia Disorders
Keywords: Hallucinations,; psychotic,; delusions,; cognitive deficits
MeSH Terms: conditions — Schizophrenia; Hallucinations; Mental Disorders; Delusions; Cognition Disorders | interventions — Single Person; 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (single and multiple doses)
- AQW051 Dose 1 (Experimental)
  Interventions: Drug: AQW051 2 mg (single and multiple doses)
- AQW051 Dose 2 (Experimental)
  Interventions: Drug: AQW051 15mg (single and multiple doses)
- AQW051 Dose 3 (Experimental)
  Interventions: Drug: AQW051 100mg (single dose), and 50mg (multiple doses)

INTERVENTIONS:
Drug: Placebo (single and multiple doses)
  Arms: Placebo
Drug: AQW051 2 mg (single and multiple doses)
  Arms: AQW051 Dose 1
Drug: AQW051 15mg (single and multiple doses)
  Arms: AQW051 Dose 2
Drug: AQW051 100mg (single dose), and 50mg (multiple doses)
  Arms: AQW051 Dose 3

SUMMARY:
This PoC study is designed to assess the cognitive effects of doses of AQW051 in patients with chronic stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia
2. Symptomatically stable and currently treated with a stable regimen for at least 3 (three) months prior to dosing with one of the following second generation of antipsychotics: risperidone, paliperidone, quetiapine, ziprasidone, aripiprazole.
3. Specific cognitive impairment
4. Smokers and non-smokers

Exclusion Criteria:

1. Current treatment with an anticholinergic or other agent known to adversely interfere with the cholinergic system, and/ or treatment with cholinesterase inhibitor within the last three (3) months prior to dosing.
2. Current treatment with conventional antipsychotics (e.g fluphenazine, haloperidol) or clozapine.
3. History of neuroleptic malignant syndrome.
4. Diagnosis of substance abuse (other than nicotine) within the last month and alcohol or substance dependence (other than nicotine) within the last 6 months.
5. Any clinically significant suicidal ideation (Type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last month) or previous history of suicide behavior Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Effects of single oral doses of AQW051 versus placebo on cognitive function as measured by selected CogState tests | 132 days Part A, 121 days Part B (screening to study completion)

SECONDARY OUTCOMES:
Effects of single oral doses of AQW051 versus placebo on cognitive function as measured by selected MATRICS Consensus Cognitive Battery (MCCB) tests | 132 days Part A, 121 days Part B (screening to study completion)
Effects of multiple oral doses of AQW051 versus placebo on cognitive function as measured by selected CogState tests and selected MCCB tests | 132 days Part A, 121 days Part B (screening to study completion)
Correlation of the cognitive domains measured by MCCB versus CogState | 132 days Part A, 121 days Part B (screening to study completion)
Pharmacokinetics, safety and tolerability of single and multiple doses of AQW051 as compared to placebo | 132 days Part A, 121 days Part B (screening to study completion)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - PAREXEL (California Clinical Trials Medical Group), 1560 Chevy Chase Drive, Suite 140,, Glendale, California
  - CRI Worldwide, 1113 Hospital Dr. Suite 202,, Willingboro, New Jersey

REFERENCES:
- See also: Results for CAQW051A2205 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12543